CLINICAL TRIAL: NCT00461526
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of TRN-002 (Crofelemer) for the Symptomatic Treatment of Diarrhea-Predominant Irritable Bowel Syndrome (d-IBS) in Females
Brief Title: Diarrhea Predominant Irritable Bowel Syndrome in Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Michelle Widmann, Associate Director, Clinical Operations, Salix Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRN-002-202
Record Dates: First submitted 2006-11-09; First posted 2007-04-18 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; d-IBS; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — crofelemer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 125 mg crofelemer (Experimental)
  Interventions: Drug: crofelemer
- placebo (Placebo Comparator)
  Interventions: Drug: crofelemer

INTERVENTIONS:
Drug: crofelemer — 125 mg crofelemer vs. placebo

SUMMARY:
Clinical Trial with TRN-002 in Women with Irritable Bowel Syndrome (IBS)

The purpose of this study is to investigate the safety and effectiveness of a new investigational drug in women for the treatment of diarrhea-predominant irritable bowel syndrome. The investigational drug is a natural product taken from a plant that grows in South America. The study medication will be administered orally twice a day. Subjects will be not able to remain on certain standard IBS medications (anti-diarrheals) while participating in the study. The total duration of the study is 18 weeks.

The study requires five study visits that include physical exams, ECG, blood draws, laboratory studies, and a colon procedure (such as a colonoscopy or flexible sigmoidoscopy if an appropriate procedure has not been performed in the last 5 years.) Participants will be asked to make entries into a touch-tone telephone diary on a daily basis.

Participants must meet all of the following criteria:

* Females at least 18 years of age
* Diagnosis of diarrhea predominant Irritable Bowel Syndrome
* Willingness to make daily calls on a touch-tone telephone
* Willingness to have an endoscopic and/or radiologic bowel evaluation, if you have not received one in the past 5 years.
* Willingness to take an approved method of birth control (if required)

Participants CANNOT meet any of the following criteria:

* Serious medical or surgical conditions
* Colon Cancer, Crohns Disease or Ulcerative Colitis
* Pregnant or breast feeding

DETAILED DESCRIPTION:
Clinical Trial with TRN-002 in Women with Irritable Bowel Syndrome (IBS)

The purpose of this study is to investigate the safety and effectiveness of a new investigational drug in women for the treatment of diarrhea-predominant irritable bowel syndrome. The investigational drug is a natural product taken from a plant that grows in South America. The study medication will be administered orally twice a day. Subjects will be not able to remain on certain standard IBS medications (anti-diarrheals) while participating in the study. The total duration of the study is 18 weeks.

The study requires five study visits that include physical exams, ECG, blood draws, laboratory studies, and a colon procedure (such as a colonoscopy or flexible sigmoidoscopy if an appropriate procedure has not been performed in the last 5 years.) Participants will be asked to make entries into a touch-tone telephone diary on a daily basis.

Participants must meet all of the following criteria:

* Females at least 18 years of age
* Diagnosis of diarrhea predominant Irritable Bowel Syndrome
* Willingness to make daily calls on a touch-tone telephone
* Willingness to have an endoscopic and/or radiologic bowel evaluation, if you have not received one in the past 5 years.
* Willingness to take an approved method of birth control (if required)

Participants CANNOT meet any of the following criteria:

* Serious medical or surgical conditions
* Colon Cancer, Crohns Disease or Ulcerative Colitis
* Pregnant or breast feeding

ELIGIBILITY:
Inclusion Criteria:

* Females at least 18 years of age
* Diagnosis of diarrhea predominant Irritable Bowel Syndrome
* Willingness to make daily calls on a touch-tone telephone
* Willingness to have an endoscopic and/or radiologic bowel evaluation, if you have not received one in the past 5 years.
* Willingness to take an approved method of birth control (if required)

Exclusion Criteria:

* Serious medical or surgical conditions
* Colon Cancer, Crohns Disease or Ulcerative Colitis
* Pregnant or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of TRN-002 when administered twice daily for 12 consecutive weeks. | March 2008
To assess the efficacy of TRN-002 when administered twice daily for 12 consecutive weeks. | March 2008

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Clinical Research Associates, LLC, Huntsville, Alabama
  - Radiant Research, Chandler, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Community Clinical Trials, Orange, California
  - Advanced Clinical Research Institute, Orange, California
  - Medical Associates Research Group, San Diego, California
  - Boulder Medical Center, PC, Boulder, Colorado
  - Rocky Mountain Gastroenterology Associates, Thornton, Colorado
  - Litchfield County Gastroenterology Associates, LLC, Torrington, Connecticut
  - Washington Gastroenterology, PC, Washington D.C., District of Columbia
  - Consultants of Clinical Research of South Florida, Boynton Beach, Florida
  - University Clinical Research - DeLand, DeLand, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Digestive and Liver Disease Consultants, PC, Clive, Iowa
  - Trover Center for Clinical Studies, Madisonville, Kentucky
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Gastroenterology Associates, Jackson, Mississippi
  - Toby Village Office Park, Pittsford, New York
  - LeBauer Research Associates, PA, Greensboro, North Carolina
  - Vital re:Search, Greensboro, North Carolina
  - Bethany Medical Center, High Point, North Carolina
  - Hanover Medical Specialist, PA, Wilmington, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Akron Gastroenterology Associates, Inc., Akron, Ohio
  - Research Solutions Corp., Cincinnati, Ohio
  - Gastrointestinal & Liver Disease Consultants, Dayton, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Grand View Medical Research, Sellersville, Pennsylvania
  - Anderson Gastroenterology Associates, LLC, Anderson, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Gastroenterology Center of the MidSouth, PC, Germantown, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - Gastroenterology Associates, Kingsport, Tennessee
  - Austin Gastroenterology, PA, Austin, Texas
  - Trinity Clinic - Corsicana, Corsicana, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Vantage Clinical Research Group, Olympia, Washington
  - Northside Internal Medicine, Spokane, Washington

REFERENCES:
- [Derived] Nee J, Salley K, Ludwig AG, Sommers T, Ballou S, Takazawa E, Duehren S, Singh P, Iturrino J, Katon J, Lee HN, Rangan V, Lembo AJ. Randomized Clinical Trial: Crofelemer Treatment in Women With Diarrhea-Predominant Irritable Bowel Syndrome. Clin Transl Gastroenterol. 2019 Dec;10(12):e00110. doi: 10.14309/ctg.0000000000000110. PMID 31800542